CLINICAL TRIAL: NCT00385398
Title: Phase II Quality of Life Study of Stereotactic RadioSurgery, Temozolomide and Erlotinib Chemotherapy for the Treatment of 1-3 Brain Metastases in Non-small Cell Lung Cancer
Brief Title: QOL-Stereotactic RadioSurgery, Temozolomide + Erlotinib-Rx of 1-3 Brain Metastases in NSCLC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding and drug supply
Sponsor: University of Medicine and Dentistry of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Schering-Plough (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030601; P30CA072720 (NIH); 0220060108 (Other: IRB Number); CINJ-NJ1506; CDR0000539474
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: tumors metastatic to brain; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Brain Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Temozolomide; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: erlotinib hydrochloride — Erlotinib will be administered orally on at a dose of 200 mg/day on Days 1-23 of each 28 day cycle.
Drug: temozolomide — Temozolomide will be administered orally at a dose of 150 mg/m2 on Days 1-5 for Cycle 1 then increased to 200 mg/m2 for Cycle 2 forward.
Radiation: stereotactic radiosurgery — Stereotactic radiosurgery will be performed prior to chemotherapy.

SUMMARY:
RATIONALE: Treatment with radiosurgery, temozolomide, and erlotinib may affect brain function (the ability to think, learn, remember, and judge) in patients with non-small cell lung cancer and brain metastases. A study that evaluates brain function may help doctors plan the best treatment.

PURPOSE: This phase II trial is studying the effect of radiosurgery, temozolomide, and erlotinib on brain function in patients with non-small cell lung cancer and brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the effect of stereotactic radiosurgery, temozolomide, and erlotinib hydrochloride on cognitive function in patients with non-small cell lung cancer and brain metastases.

Secondary

* Determine the feasibility and safety of this regimen, in terms of tumor response, time to tumor progression in brain, survival, physical functioning, and quality of life, in these patients.
* Determine the frequency of O6-methylguanine-DNA methyltransferase promoter methylation in these patients.

OUTLINE: This is a multicenter study.

Patients undergo stereotactic radiosurgery on day -7. Patients receive oral temozolomide once daily on days 1-5 and oral erlotinib hydrochloride once daily on days 1-23. Treatment with temozolomide and erlotinib hydrochloride repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo cognitive function evaluation as measured by Mini-Mental Status Exam administration and scoring; quality of life assessment as measured by Functional Assessment of Cancer Therapy subscale; and physical functioning assessment as measured by Katz index of activities of daily living and Karnofsky performance status at baseline and then every 8 weeks during study treatment.

Tumor tissue is examined by O6-methylguanine-DNA methyltransferase (MGMT gene) promotor methylation.

After completion of study therapy, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 54 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed non-small cell lung cancer meeting the following criteria:

  * One to 3 brain metastases, meeting the following criteria:

    * No larger than 3 cm
    * Greater than 5 mm from the optic apparatus
    * Not involving the brainstem, pons, medulla, or midbrain
  * Stable systemic disease for the past 3 months

    * Less than 3 months since completion of primary treatment
* Measurable CNS disease as defined by RECIST criteria
* No leptomeningeal disease documented by MRI or cerebrospinal fluid cytologic evaluation

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 12 weeks
* Karnofsky performance status 60-100%
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10 g/dL
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST ≤ 3.0 times ULN
* Serum creatinine ≤ 1.5 mg/dL
* Creatinine clearance > 50 mL/min
* No other malignancy within the past 5 years, except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No concurrent major medical illness or psychiatric impairment that, in the investigator's opinion, would preclude study participation
* No concurrent active infections
* No known HIV positivity
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception during and for 3 months after completion of study treatment

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior complete resection of all brain metastases
* No prior brain radiation therapy
* No prior temozolomide or erlotinib hydrochloride
* No concurrent enzyme-inducing anti-epileptic drugs
* No concurrent recombinant interleukin-11
* No other concurrent anticancer investigational or commercial agents or therapies, including chemotherapy, immunotherapy, hormonal cancer therapy, radiation therapy, or cancer surgery
* No concurrent enrollment on another clinical trial
* Surgery for symptomatic brain lesions prior to radiosurgery allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 2 years

SECONDARY OUTCOMES:
Tumor response | 2 years
Time to tumor progression in brain | 2 years
Survival | 2 years
Quality of life as measured by FACT subscale | 2 years
Physical functioning as measured by Karnofsky performance status and Katz index of activities of daily living | 2 years
Frequency of O6-methylguanine-DNA methyltransferase promoter methylation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Molly Gabel, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey